CLINICAL TRIAL: NCT00073151
Title: A Phase II Study of ABT-751 in Patients With Non-Small Cell Lung Cancer Refractory to Taxane Regimens
Brief Title: A Study of ABT-751 in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-448; NCT00080730 (obsolete NCT alias)
Record Dates: First submitted 2003-11-17; First posted 2003-11-18 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ABT751

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABT-751

SUMMARY:
The purpose of the study is to determine if ABT-751 will decrease tumors, and determine how long the tumor shrinkage can be maintained in patients with non-small cell lung cancer. Patients will receive ABT-751 by mouth daily for 21 days. Patients will be off drug for 7 days before starting the next cycle of drug.

ELIGIBILITY:
Inclusion Criteria

* Stage IIIB or IV non-small cell lung cancer.
* Recurrent tumor following treatment with paclitaxel or docetaxel.
* Able to tolerate normal activities of daily living.
* Adequate bone marrow, kidney and liver function.

Exclusion Criteria

* Pregnant or breast feeding.
* Anti-tumor therapy within 4 weeks of the start of ABT-751 administration.
* CNS metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-09; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate in subjects with NSCLC | 1 year

SECONDARY OUTCOMES:
Time to Tumor Progression (TTP) | 1 year
Survival | 2 years
Toxicities associated with treatment administration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Eliopoulos, MD, Study Director — Abbott
Locations (17):
- United States (17):
  - Oncology Hematology Group of South Florida, Miami, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Maryland Greenbaum Cancer Center, Baltimore, Maryland
  - Oncology & Hematology Associates of Kansas City, PA, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Regional Cancer Center, Albany, New York
  - Raleigh Hematology Oncology, Cary, North Carolina
  - Dayton Oncology and Hematology, Kettering, Ohio
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - West Cancer Clinic, Memphis, Tennessee
  - Texas Oncology, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - Cancer Care Northwest, Spokane, Washington
  - Northwest Cancer Specialists, Vancouver, Washington
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin